CLINICAL TRIAL: NCT05825794
Title: Active Pharmacovigilance of Anti-cancer Medicines in Pediatric and Young Adult Patients.
Brief Title: Active Pharmacovigilance of Anti-cancer Medicines
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: IRCCS Burlo Garofolo (Other)
Responsible Party: Sponsor
Other Study IDs: AIFA FVG 2019
Record Dates: First submitted 2023-03-29; First posted 2023-04-24 (Actual); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Oncology; Drugs; Pharmacovigilance
Keywords: Oncology; Drugs; Active pharmacovigilance
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Pharmacovigilance (PV), defined by the World Health Organization (WHO) as the "science and activities related to the detection, evaluation, understanding and prevention of adverse effects or any other drug-related problem", aims to improve patient safety and quality of life. There are several objectives of PV, starting with the collection and management of safety data, to promote the safe and effective use of medicines. PV also aims to provide information on drug safety to health professionals and patients, and it contributes to updating drug labels. Finally, it is active in risk management, risk minimization and the prevention of adverse effects and other drug-related problems. As defined by WHO, an adverse event (AE) is "any untoward medical occurrence that may be present during treatment with a medicine, but which does not necessarily have a causal relationship with this treatment". When there is a causal relationship with the treatment, an AE is classified as an adverse drug reaction (ADR). The collection and reporting of AEs is a process that starts from the drug development phase and proceeds continuously throughout the life cycle of the drug, and it aims to assess the benefits-to-toxicity ratios (in other words, the safety and efficacy) of all medicines. Reports of ADRs must accurately describe the case and be meaningful to health professionals worldwide. The aim of this project is to evaluate the impact of an active prescription surveillance of anti-cancer drugs carried out by the clinical pharmacist in pediatrics and young adults.

ELIGIBILITY:
Inclusion Criteria:

* patients aged <25 years;
* receiving cytotoxic, targeted-therapy, immunotherapy drugs for the treatment of solid and hematologic cancers
* giving consent to study participation

Exclusion Criteria:

* presence of cognitive problems

Max Age: 25 Years | Sex: All
Age Groups: Child, Adult
Study Population: Pediatric and young adult patients requiring the administration of anticancer drugs
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-10-28 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
To quantify the number of grade 3-5 ADRs reported during the active surveillance period | Through study completion, an average of 3 years
  ADRs grades will be standardized using the Common Terminology Criteria for Adverse Events (CTCAE) v4.3.
To compare the number of grade 3-5 ADRs reported during the active surveillance period with the number of grade 3-5 ADRs reported in the previous years | Through study completion, an average of 3 years
  Period of equal length will be compared

CONTACTS AND LOCATIONS:
Overall Officials: Marta Trojniak, PharmD, Principal Investigator — IRCCS materno infantile Burlo Garofolo
Locations (1):
- IRCCS materno infantile Burlo Garofolo, Trieste, Italy